CLINICAL TRIAL: NCT01335204
Title: Phase Ib/IIa Study of Cabazitaxel Plus Bavituximab for Patients With Castration-resistant Prostate Cancer Previously Treated With Chemotherapy
Brief Title: Ph Ib/IIa Study of Cabazitaxel Plus Bavituximab in Castration-resistant Prostate Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: lack of funding
Sponsor: Medical University of South Carolina (Other)
Collaborators: Peregrine Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MUSC 101637; HS#2011-8083 (Other: University of California, Irvine); NCI-2011-01248 (Other: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2011-04-11; First posted 2011-04-14 (Estimated); Results first posted 2018-07-13 (Actual); Last update posted 2018-07-13 (Actual); Status verified 2018-06

CONDITIONS: Prostate Cancer; Prostatic Neoplasms
Keywords: Castration-resistant prostate cancer; Prostate Cancer; JEVTANA; Cabazitaxel; Bavituximab
MeSH Terms: conditions — Prostatic Neoplasms | interventions — cabazitaxel; bavituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cabazitaxel plus bavituximab (Experimental): Cabazitaxel (25 mg/m2) will be administered IV on Day 1 of each 21-day treatment cycle. Bavituximab (3 mg/kg) will be administered as an IV infusion on a weekly basis (Cycle 1 Day 2, all other cycles Day 1; day 8; day 15) for 8 cycles.
  Interventions: Drug: Cabazitaxel plus bavituximab

INTERVENTIONS:
Drug: Cabazitaxel plus bavituximab — Cabazitaxel (25 mg/m2) will be administered IV on Day 1 of each 21-day treatment cycle, and bavituximab (3 mg/kg) will be administered as an IV infusion on a weekly basis (Cycle 1 Day 2, all other cycles Day 1; day 8; day 15) for 8 cycles.
  Other Names: JEVTANA® (cabazitaxel)

SUMMARY:
This is a Phase Ib/IIa Study of Cabazitaxel plus Bavituximab in patients with castration-resistant prostate cancer (CRPC). The current study is designed to determine if the addition of bavituximab to cabazitaxel will improve progression free survival (PFS) or overall survival (OS). In addition, the Lead Researcher is requiring the collection of urine, and blood specimens for future research.

This study will enroll patients with CRPC, who have been previously treated with docetaxel or a docetaxel-containing regimen. Patients may be intolerant of, or resistant to, docetaxel, or may have been previously treated with the agent without definite disease progression during therapy.

Patients must meet the study eligibility criteria and must be competent to give informed consent.

DETAILED DESCRIPTION:
Cabazitaxel will be administered IV on day 1 of each 21-day treatment cycle. Bavituximab (3 mg/kg) will be administered as an intravenous (IV) infusion on a weekly basis (Cycle 1 Day 2, all other cycles Day 1; day 8, day 15). Patients will receive cabazitaxel (day 1) plus bavituximab weekly of each 21-day cycle for up to 8 cycles.

Up to 31 patients will be enrolled to ensure 28 evaluable subjects. The accrual period is expected to be between 12 to 18 months (1-1.5 years).

Subjects will remain on the treatment phase of the study until any of the following events occur:

* Disease progression as evidenced by an increase in the prostate-specific antigen (PSA) level, worsening of pain, or disease progression by Response Evaluation Criteria in Solid Tumors (RECIST)
* Completion of 8 cycles of cabazitaxel-bavituximab therapy (day 169)
* Development of toxicity that, in the investigator's judgment, precludes further study participation
* Significant protocol violations or noncompliance on the part of the patient or investigator
* The investigator's judgment that discontinuation is in the patient's best interest
* Initiation of alternative antineoplastic treatments.
* Refusal of the patient to continue treatment or follow-up
* Loss to follow-up

After completion of the treatment phase, subjects will remain on the followup phase of the study until any of the following events occur:

* Refusal of the patient to continue treatment or follow-up
* Loss to follow-up
* Death
* The investigator's judgment that discontinuation is in the patient's best interest

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent has been obtained.
* Adults 18 years of age or older with a life expectancy of at least 3 months.
* Histologically confirmed castration-resistant prostate cancer (CRPC). Patient must have demonstrated a rising PSA level above the androgen-deprivation therapy (ADT) nadir, on at least two determinations four weeks or more apart. ADT is defined as treatment with a Luteinizing-hormone-releasing hormone (LHRH) agonist or orchiectomy.
* Treatment with only one prior chemotherapy regimen, which must contain docetaxel as a single agent or in combination with other agents. Patients may be intolerant of, or resistant to, the cytotoxic drug combination.
* Patients on ADT must be willing to continue ADT for the duration of their participation in this protocol. ADT cannot be initiated, and ADT dose/agents may not be changed during the study.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
* Adequate hematologic function (absolute neutrophil count [ANC] ≥ 1,500 cells/μL; hemoglobin ≥ 8 g/dL, platelets ≥ 100,000/μL).
* Adequate renal function (serum creatinine ≤ 1.5 mg/dL or calculated creatinine clearance ≥ 60 mL/min).
* Adequate hepatic function (bilirubin ≤ 1.0 x upper limit of normal [ULN], alanine aminotransferase [ALT] ≤ 1.5 x ULN, aspartate aminotransferase [AST] ≤ 1.5 x ULN).
* Prothrombin time (PT) / international normalized ratio (INR) ≤ 1.5 × ULN.
* Activated partial thromboplastin (aPTT) time ≤ 1.5 × ULN.
* Prostate-specific antigen (PSA) level of at least 2 ng/mL.
* New York Heart Association classification I or II.
* All patients of reproductive potential must agree to use an approved form of contraception (as determined by the investigator).

Exclusion Criteria:

* Known history of bleeding diathesis or coagulopathy (e.g., von Willebrand disease or hemophilia).
* Any history of thromboembolic events (e.g., deep vein thrombosis or pulmonary thromboembolism); central venous catheter-related thrombosis > 6 months before Screening is allowed.
* Ongoing therapy with oral or parenteral anticoagulants; patients on low-dose anticoagulants to maintain patency of central venous catheters are eligible.
* Grade 2 or higher peripheral neuropathy (e.g., numbness, tingling, and/or pain in distal extremities).
* Radiotherapy (teletherapy or brachytherapy) , chemotherapy or estrogen agonist within 28 days before Study Day 1.
* Systemic radiotherapy (Sm-153, Sr-89) within 56 days before study day 1.
* Symptomatic or clinically active brain metastases.
* Major surgery within 28 days of Study Day 1.
* Uncontrolled intercurrent disease (eg, diabetes, hypertension, thyroid disease).
* Any history of cerebrovascular accident, or transient ischemic attack at any time, or history of symptomatic coronary artery disease < 6 months before screening.
* A history of any condition requiring anti-platelet therapy (eg, phosphodiesterase inhibitors, adenosine diphosphate receptor antagonists), with the exception of general cardiovascular prophylaxis with aspirin (≤ 325 mg/day).
* Serious non-healing wound (including wound healing by secondary intention, ulcer, or bone fracture).
* Known chronic infection with human immunodeficiency virus (HIV) or viral hepatitis.
* Contraindication to intravenous (IV) contrast media.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2011-06; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Lilly, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cabazitaxel Plus Bavituximab
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cabazitaxel Plus Bavituximab
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Probability of Progression-free Survival at Day 85
Description: The primary objective of this study is to determine the probability of progression-free survival (PFS) after 12 weeks of therapy in subjects with CRPC treated with cabazitaxel + bavituximab.
Time Frame: 12 weeks
Population: This study terminated early, so outcomes were not analyzed.
Arm/Group | Cabazitaxel Plus Bavituximab
Number analyzed (Participants) | 0

2. Secondary Outcome: Measurement of PSA Response Rate
Description: To estimate the PSA response rate from cabazitaxel + bavituximab therapy in CRPC patients previously treated with docetaxel. PSA response rate will be assessed at multiple time points during the 24 wks of study treatment.
Time Frame: 24 weeks
Population: This study terminated early, so outcomes were not analyzed.
Arm/Group | Cabazitaxel Plus Bavituximab
Number analyzed (Participants) | 0

3. Secondary Outcome: Objective Response Rate by RECIST for Patients With Measurable Disease
Description: To estimate the objective response rate from cabazitaxel + bavituximab therapy in CRPC patients previously treated with docetaxel. Objective response rate will be assessed at day 85, 169
Time Frame: 24 weeks
Population: This study terminated early, so outcomes were not analyzed.
Arm/Group | Cabazitaxel Plus Bavituximab
Number analyzed (Participants) | 0

4. Secondary Outcome: Overall Survival
Description: To estimate the overall survival in subjects with CRPC (previously treated with docetaxel) following cabazitaxel + bavituximab therapy. Overall survival will be assessed continually during the duration of the study.
Time Frame: 24+ weeks
Population: This study terminated early, so outcomes were not analyzed.
Arm/Group | Cabazitaxel Plus Bavituximab
Number analyzed (Participants) | 0

5. Secondary Outcome: Number of With Grade 3 or 4 Toxicities
Description: To document the toxicity of cabazitaxel + bavituximab therapy in CRPC patients previously treated with docetaxel. Toxicity will be assessed continually during the 24 wks of study therapy.
Time Frame: 24 weeks
Measure: Number; unit: grade 3 or 4 toxicities
Arm/Group | Cabazitaxel Plus Bavituximab
Number analyzed (Participants) | 4
grade 3 or 4 toxicities | 5

6. Secondary Outcome: Progression-free Survival (PFS)
Description: Determination of progression-free survival in subjects treated with cabazitaxel + bavituximab for CRPC previously treated with docetaxel. PFS will be assessed continually during the entire study.
Time Frame: 24+ weeks
Population: This study terminated early, so outcomes were not analyzed.
Arm/Group | Cabazitaxel Plus Bavituximab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Cabazitaxel Plus Bavituximab
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 4/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cabazitaxel Plus Bavituximab (N=4)
anemia (Blood and lymphatic system disorders) | 1 (1)
febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
fatigue (General disorders) | 2 (2)
neutrophil count decrease (Investigations) | 2 (2)
chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
headache (Nervous system disorders) | 1 (1)
memory impairment (Nervous system disorders) | 1 (1)
peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
diarrhea (Gastrointestinal disorders) | 1 (1)
oral pain (Gastrointestinal disorders) | 1 (1)
stomach pain (Gastrointestinal disorders) | 1 (1)
vomiting (Gastrointestinal disorders) | 1 (1)
anorexia (Metabolism and nutrition disorders) | 1 (1)
hematuria (Renal and urinary disorders) | 1 (1)
urinary urgency (Renal and urinary disorders) | 1 (1)
alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
hypertension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes